CLINICAL TRIAL: NCT04630067
Title: A Phase Ia/b Randomized, Single-blinded, Placebo-controlled Study to Evaluate the Safety, Tolerability, Immunogenicity, and Pharmacokinetics of Single Ascending Doses of AZD3427 in Healthy Volunteers and Multiple Ascending Doses of AZD3427 in Patients With Heart Failure (HFrEF and HF With EF ≥ 41%)
Brief Title: Assessment of Safety, Tolerability, Immunogenicity, and Pharmacokinetics of AZD3427
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D8330C00001
Record Dates: First submitted 2020-10-27; First posted 2020-11-16 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure
Keywords: Heart failure with reduced ejection fraction; Heart failure with ejection fraction of ≥ 41%; AZD3427; First-time-in-human
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- AZD3427: Cohort 1a (Experimental): Participants will receive single SC dose A of AZD3427 on Day 1.
  Interventions: Drug: AZD3427
- AZD3427: Cohort 2a (Experimental): Participants will receive single SC dose B of AZD3427 on Day 1.
  Interventions: Drug: AZD3427
- AZD3427: Cohort 3a (Experimental): Participants will receive single SC dose C of AZD3427 on Day 1.
  Interventions: Drug: AZD3427
- AZD3427: Cohort 4a (Experimental): Participants will receive single SC dose D of AZD3427 on Day 1.
  Interventions: Drug: AZD3427
- AZD3427: Cohort 5a (Experimental): Participants will receive single IV dose E of AZD3427 on Day 1.
  Interventions: Drug: AZD3427
- AZD3427: Cohort 6a (Experimental): Participants of Japanese descent will receive single SC dose anticipated equal to the highest dose of AZD3427 in the global cohorts on Day 1.
  Interventions: Drug: AZD3427
- AZD3427: Cohort 7a (Experimental): Participants will receive single SC dose F of AZD3427 on Day 1
  Interventions: Drug: AZD3427
- Part A: Placebo (Placebo Comparator): Participants will receive single SC or IV dose of placebo matched to AZD3427 on Day 1.
  Interventions: Drug: Placebo
- AZD3427: Cohort 1b (Experimental): Participants with HFrEF will receive SC dose A of AZD3427 on Days 1, 8, 15, 22, and 29.
  Interventions: Drug: AZD3427
- AZD3427: Cohort 2b (Experimental): Participants with HF with EF ≥ 41% will receive SC dose A of AZD3427 on Days 1, 8, 15, 22, and 29.
  Interventions: Drug: AZD3427
- AZD3427: Cohort 3b (Experimental): Participants with HFrEF will receive SC dose B of AZD3427 on Days 1, 8, 15, 22, and 29.
  Interventions: Drug: AZD3427
- AZD3427: Cohort 4b (Experimental): Participants with HF with EF ≥ 41% will receive SC dose B of AZD3427 on Days 1, 8, 15, 22, and 29.
  Interventions: Drug: AZD3427
- AZD3427: Cohort 5b (Experimental): Participants with HFrEF will receive SC dose C of AZD3427 on Days 1, 8, 15, 22, and 29.
  Interventions: Drug: AZD3427
- AZD3427: Cohort 6b (Experimental): Participants with HF with EF ≥ 41% will receive SC dose C of AZD3427 on Days 1, 8, 15, 22, and 29.
  Interventions: Drug: AZD3427
- Part B: Placebo (Placebo Comparator): Participants with HFrEF or HF with EF ≥ 41% will receive SC dose of placebo matched to AZD3427 on Days 1, 8, 15, 22, and 29.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD3427 — Participants will receive SC or IV dose of AZD3427 as per the arm they are randomized.
  Arms: AZD3427: Cohort 1a; AZD3427: Cohort 1b; AZD3427: Cohort 2a; AZD3427: Cohort 2b; AZD3427: Cohort 3a; AZD3427: Cohort 3b; AZD3427: Cohort 4a; AZD3427: Cohort 4b; AZD3427: Cohort 5a; AZD3427: Cohort 5b; AZD3427: Cohort 6a; AZD3427: Cohort 6b; AZD3427: Cohort 7a
Drug: Placebo — Participants will receive SC or IV dose of placebo matched to AZD3427 as per the arm they are randomized.
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
This first-time-in-human (FTIH) study will be conducted to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of single doses of AZD3427 in healthy volunteers and multiple doses of AZD3427 in patients with heart failure (HF).

DETAILED DESCRIPTION:
This is a multi-center single and multiple ascending dose study (SAD and MAD).

Part A (SAD) will include 7 cohorts (8 healthy volunteers in each cohort) and will randomize to AZD3427 or placebo, in a 6:2 ratio. One cohort will entirely include participants of Japanese descent.

Part B (MAD) will include 6 cohorts (8 heart failure patients in each cohort) and will randomize to AZD3427 or placebo in a 6:2 ratio. Of these, 3 cohorts will contain participants with heart failure with reduced ejection fraction [HFrEF] and the other 3 cohorts will comprise of participants with heart failure with HF with ejection fraction (EF) ≥ 41%. There will be a maximum screening period of 27 days. Participants in part A and B will undergo study drug administration on Day 1. In addition, participants in part B will return for 4 additional doses on Days 8, 15, 22, and 29. Participants will be followed for at least 50 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Part A will include healthy men and non-pregnant, non-lactating females of non-childbearing potential with a body mass index (BMI) of 18-30 kg/m^2 and a weight of 55-100 kg. One cohort will require participants be of Japanese descent
* Part B will include men and non-pregnant, non-lactating females of non-childbearing potential
* Participants have a BMI of 18-40 kg/m^2 and a weight of 55-136 kg
* Participants with a diagnosis of stage C HF New York Heart Association (NYHA) Class I-III on stable medical therapy for at least 12 weeks
* Participants with diagnosis of HFrEF will be defined as those with EF ≤ 40% and HF with EF ≥ 41%
* Participants either with N-terminal prohormone of brain natriuretic peptide (NT-proBNP) > 125 pg/mL or BNP > 35 pg/mL (46)

Exclusion Criteria:

Both Part A and Part B will exclude participants with any of the following:

* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of study drug or planned surgical procedure before study completion
* History of vascular and left ventricular aneurysms or prior dissections
* Any history of joint hypermobility, Marfan's syndrome, or any connective tissue disorder
* Clinical signs and symptoms consistent with Coronavirus disease-19 or confirmed infection within the last 4 weeks
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity injection devices or to drugs with a similar chemical structure or class to AZD3427 or any component of AZD3427

In addition, Part A will exclude participants with any of the following:

* Alanine Aminotransferase (ALT) > Upper limit of normal (ULN)
* Aspartate Aminotransferase (AST) > ULN
* Total bilirubin > ULN (unless due to Gilbert's syndrome)
* Creatinine > ULN
* White blood cell (WBC) count < Lower limit of normal (LLN)
* Hemoglobin < LLN
* Prolonged QTcF > 450 m
* Shortened QTcF < 340 ms
* Family history of long QT syndrome
* PR (PQ) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation)
* PR (PQ) interval prolongation (> 240 ms) intermittent second (Wenckebach block while asleep is not exclusive) or third-degree atrioventricular (AV) block, or AV dissociation
* Persistent or intermittent complete bundle branch block, incomplete bundle branch block, or intraventricular conduction delay with QRS > 110 ms. Participants with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of eg, ventricular hypertrophy or pre-excitation

In addition, Part B will exclude participants with any of the following:

* Atrial fibrillation or flutter occurring in the past year
* Clinically significant ventricular arrhythmias under treatment
* High-degree AV block II-III or sinus node dysfunction
* Implanted permanent pacemaker or implantable cardioverter defibrillator for which the participant is pacing-dependent
* Severe right-sided valvular heart disease; severe mitral regurgitation; moderate or severe mitral stenosis, severe aortic regurgitation and mild, moderate or severe aortic stenosis
* Other conditions where vasodilatory therapy may be contraindicated (hypertrophic obstructive cardiomyopathy, and restrictive cardiomyopathy)
* Congenital heart disease
* NYHA HF Class IV
* Occurrence in the last 6 months of acute coronary syndrome, percutaneous coronary intervention, cerebrovascular accident or transient ischemic attack, HF hospitalization; history or suspicion of cardiac amyloidosis
* ALT > 1.5 × ULN
* AST > 1.5 × ULN
* Total bilirubin > ULN (unless due to Gilbert's syndrome)
* Impaired renal function, defined as eGFR < 30 mL/min/1.73m^2 assessed by the Chronic Kidney Disease Epidemiology Collaboration equation
* WBC < LLN
* Hemoglobin < 10g/L
* PR (PQ) interval prolongation (> 220 ms)
* Participants with persistent BBB and QRS (ECG interval measured from the onset of the QRS complex to the J point) duration > 130 ms. Participants with intraventricular conduction delay and QRS duration < 130 ms

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events and Serious Adverse Events | Part A: Day 1 until Day 50 or Early termination visit (E/T); Part B: Day 1 until Day 78 or E/T
  Assessment of the safety and tolerability of single and multiple ascending doses of AZD3427.

SECONDARY OUTCOMES:
Maximum Observed Serum (peak) Drug Concentration (Cmax) of AZD3427 | Part A: Day 1 (pre-dose, and 10 minutes [only for cohort 5a], 4hrs and 12hrs post-dose, and days 2, 3, 5, 8, 15, 29, and Day 50 or E/T ; Part B: Day 1 (Pre-dose and post-dose), days 8, 15, 22, and 29 (pre-dose); and days 2, 3, 32, 57, 71 and 78 or E/T
  Evaluation of the PK of single and multiple ascending doses of AZD3427.
Area Under the Serum Concentration-time Curve from Zero to the Last Quantifiable Concentration (AUClast) | Part A: Day 1 (pre-dose, and 10 minutes [only for cohort 5a], 4hrs and 12hrs post-dose, and days 2, 3, 5, 8, 15, 29, and Day 50 or E/T ; Part B: Day 1 (Pre-dose and post-dose), days 8, 15, 22, and 29 (pre-dose); and days 2, 3, 32, 57, 71 and 78 or E/T
  Evaluation of the PK of single and multiple ascending doses of AZD3427.
Area Under Serum Concentration-time Curve From Zero to Infinity (AUCinf) | Part A: Day 1 (pre-dose, and 10 minutes [only for cohort 5a], 4hrs and 12hrs post-dose, and days 2, 3, 5, 8, 15, 29, and Day 50 or E/T ; Part B: Day 1 (Pre-dose and post-dose), days 8, 15, 22, and 29 (pre-dose); and days 2, 3, 32, 57, 71 and 78 or E/T
  Evaluation of the PK of single and multiple ascending doses of AZD3427.
Area Under the Serum Concentration-time Curve from Zero to 168 Hours Post-dose Administration (AUC0-168) | Part A: Day 1 (pre-dose, and 10 minutes [only for cohort 5a], 4hrs and 12hrs post-dose, and days 2, 3, 5, 8, 15, 29, and Day 50 or E/T ; Part B: Day 1 (Pre-dose and post-dose), days 8, 15, 22, and 29 (pre-dose); and days 2, 3, 32, 57, 71 and 78 or E/T
  Evaluation of the PK of single and multiple ascending doses of AZD3427.
Time to Reach Peak or Maximum Observed Concentration or Response Following Drug Administration (tmax) | Part A: Day 1 (pre-dose, and 10 minutes [only for cohort 5a], 4hrs and 12hrs post-dose, and days 2, 3, 5, 8, 15, 29, and Day 50 or E/T ; Part B: Day 1 (Pre-dose and post-dose), days 8, 15, 22, and 29 (pre-dose); and days 2, 3, 32, 57, 71 and 78 or E/T
  Evaluation of the PK of single and multiple ascending doses of AZD3427.
Half-life Associated with Terminal Slope (λz) of a Semi-logarithmic Concentration-time Curve (t½λz) | Part A: Day 1 (pre-dose, and 10 minutes [only for cohort 5a], 4hrs and 12hrs post-dose, and days 2, 3, 5, 8, 15, 29, and Day 50 or E/T ; Part B: Day 1 (Pre-dose and post-dose), days 8, 15, 22, and 29 (pre-dose); and days 2, 3, 32, 57, 71 and 78 or E/T
  Evaluation of the PK of single and multiple ascending doses of AZD3427.
Number of Participants Testing Positive for the Presence of Anti-drug Antibodies (ADA) and Neutralizing Antibodies (NAb) to AZD3427 | Part A: Day 1 (pre-dose), Days 15, 29, and 50 or E/T; Part B: Days 1, 15, 29 (Pre-dose), Days 57 and 78 or E/T
  Evaluation of the immunogenicity of single and multiple ascending doses of AZD3427.
Evaluation of Positive Anti-drug Antibodies Titer | Part A: Day 1 (pre-dose), Days 15, 29, and 50 or E/T; Part B: Days 1, 15, 29 (Pre-dose), Days 57 and 78 or E/T
  Evaluation of the immunogenicity of single and multiple ascending doses of AZD3427.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, MD, Principal Investigator — Parexel Early Phase Clinical Unit (Baltimore), Harbor Hospital, 3001 S. Hanover St., Baltimore, MD 21225, United States of America (USA); David Lanfear, MD, Principal Investigator — Henry Ford Hospital, USA, MI
Locations (10):
- United States (10):
  - Research Site, Little Rock, Arkansas
  - Research Site, Glendale, California
  - Research Site, Daytona Beach, Florida
  - Research Site, Doral, Florida
  - Research Site, Hallandale, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Owensboro, Kentucky
  - Research Site, Brooklyn, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Connolly K, George R, Omar S, Matsson E, Astrand M, Althage M, Pettersen D, Mohamed E, Fang K, Lima JAC, Kujacic M, Odesjo H, Turton M, Johannesson P, Gabrielsen A, Ufnal M. Novel Relaxin Receptor RXFP1 Agonist AZD3427 in the Treatment of Heart Failure: A Phase 1a/b, First-in-Human, Randomized, Single-Blind, Placebo-Controlled Study. J Am Heart Assoc. 2024 Aug 6;13(15):e034067. doi: 10.1161/JAHA.123.034067. Epub 2024 Jul 26. PMID 39056338